CLINICAL TRIAL: NCT04031911
Title: Study of the Benefits of a Short Spa Treatment on the Elimination of Residual Lithic Fragments After Treatment
Acronym: LITHUTHERM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment due to covid 19
Sponsor: GUILLEMIN Francis, MD (Other)
Collaborators: Association Francaise pour la Recherche Thermale (Other); Conseil National des Etablissements Thermaux (Unknown)
Responsible Party: Sponsor-Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A00570-55 LITHUTHERM
Record Dates: First submitted 2019-07-17; First posted 2019-07-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Calculi, Urinary
Keywords: Urinary lithiasis; Urological treatments; Spa treatment; Posturotherapy; Lumbar percussions; Hyperdiuresis
MeSH Terms: conditions — Urinary Calculi; Urolithiasis

STUDY DESIGN:
Intervention Model Description: This clinical study will be organized in 2 arms:
  * Control group benefiting from standard support (AFU (Association Française d'Urologie) information sheet), but applied in a more supervised way (communication document, process studies, etc.).
  * Study group benefiting from a short spa treatment (5 days) with hydroposturotherapy ("HPT" arm) in Vittel or Capvern: posturotherapy, lumbar percussion and controlled hyperdiuresis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Control group benefiting from standard support (AFU (Association Française d'Urologie) information sheet), but applied in a more supervised way (communication document, process studies, etc.).
  Interventions: Device: Standard support in urology
- Study group (Experimental): Study group benefiting from a short spa treatment (5 days) with hydroposturotherapy ("HPT" arm) in Vittel or Capvern: posturotherapy, lumbar percussion and controlled hyperdiuresis.
  Interventions: Device: Hydroposturotherapy

INTERVENTIONS:
Device: Hydroposturotherapy — Hydroposturotherapy combines:
  * posturotherapy (patient placed upside down with water jets sent to the kidneys)
  * lumbar percussion
  * hyperdiuresis: prescribed quantities of water to be absorbed by the patient
  Arms: Study group
Device: Standard support in urology — Dispensing of AFU plugs Dietary advice
  Arms: Control group

SUMMARY:
Current urological therapeutic modalities are represented by extracorporeal lithotripsy (ECL), rigid (URS) or flexible (URSsple) uretero-renoscopy and percutaneous nephrolithotomy (PCNL).

They make it possible to extract the vast majority of stones by minimally invasive techniques but leave behind small residual lithic fragments (FR) that can always cause pain, infection, or promote the development of a larger stone.

A non-invasive technique that can help eliminate them would be of great benefit to many patients by avoiding painful recurrences and limiting reprocessing; combined with appropriate medical management, it would limit the rate of remote recurrences and long-term complications.

The treatment called "hydro-posturotherapy" has been developed in some spas that are approved for kidney diseases such as Vittel or Capvern. It includes several modalities: posturotherapy, lumbar percussion and hyperdiuresis.

The main objective is to compare at 3 months, on the unprepared abdomen (ASP) and the low-dose scanner without injection, the elimination of kidney stone fragments under the effect of a short spa treatment with posturotherapy, lumbar percussion and controlled hyperdiuresis compared to the recommended standard treatment. The result will be assessed in 3 categories: complete elimination (SF: "without fragments" or "stone-free"), elimination of more than 50% of the fragments; elimination of less than 50% of the fragments.

DETAILED DESCRIPTION:
Randomized multicenter controlled clinical trial comparing hydroposturotherapy in short thermal cure with standard hyperdiuresis in patients with residual stones, especially lower caliciels after urological treatment.

5 inclusion centres

* Central Hospital, Nancy
* Nancy Urology Center
* Clinique de la Croix du Sud in Toulouse
* Edouard Herriot Hospital in Lyon

The radiological images will be reviewed by the radiology department of the Central Hospital, Nancy.

ELIGIBILITY:
Inclusion Criteria:

* Major patients with urinary stones who have received minimally invasive urological treatment: extracorporeal lithotripsy (ECL), flexible uretero-renoscopy (URSsple) and percutaneous nephrolithotomy (NLPC).
* Patients with kidney stones less than 4 mm in size who are not receiving minimally invasive therapy.
* Evaluation of the number, size / volume and location of calculations by ASP & TDM low-dose, without post-operative injection.
* Information and signature of informed consent.

Exclusion Criteria:

* Patients refusing a spa treatment
* Contraindications to PTH: morbid obesity, unbalanced hypertension, pregnancy, respiratory failure, dizziness, vascular and/or ocular disorders, poly-mediated unbalanced cardiovascular pathology, orthostatic hypotension, general condition of the patient incompatible with the treatment
* Patients with Cacchi Ricci disease
* Person under the protection of justice, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Rate of SF patients (without fragment / stone free) in each arm, on the scanner and on the ASP. | 3 months after the patient's urological management
  Estimate of the rate of patients for whom all fragments have been eliminated

SECONDARY OUTCOMES:
Size of residual fragments in the cavities of the treated kidney at 3 months. | 3 months after the patient's urological management
  The size of the residual fragments will be measured in millimetres
Number of participants with complications related to residual stones or their evacuation | At inclusion, 1 month after inclusion, 3 months after inclusion
  Complications may include renal colic, low back pain, urinary tract infections
Quality of life questionnaire SF 36 : The Short Form (36) Health Survey | At inclusion, 1 month after inclusion, 3 months after inclusion
  The SF 36 questionnaire is a questionnaire measuring quality of life with 36 items grouped into 8 scales: physical activity, limitation/physical state, physical pain, perceived health, vitality, life/relationships, psychological health, limitation/psychological state
  The SF-36 is not suitable for producing an overall summary score. Indeed, the information in the individual responses is lost in the total score of the scale (since the total score can be obtained in different ways from the individual responses of the items). The recommended rating system for SF-36 is a Likert weighted system for each item. The items in the subscales are totalled to obtain a summary score for each subscale or dimension. Each of the 8 summary scores is linearly transformed on a scale from 0 (negative for health) to 100 (positive for health) to obtain a score for each subscale.
Number of intercurrent events | At inclusion, 1 month after inclusion, 3 months after inclusion
  renal colic, infection, hematuria), work stoppages, medical prescriptions, hospitalizations, urological procedures.
Medico-economic study of the benefit of the thermal cure | 3 months after inclusion of patients in the cure group
  Study of the benefits of hydroposturotherapy in terms of avoided management costs

CONTACTS AND LOCATIONS:
Overall Officials: Jacques HUBERT, PH, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU, Nancy, France

IPD SHARING:
Plan to Share IPD: No